CLINICAL TRIAL: NCT04913415
Title: Study to Evaluate a Low Suction (LS) Versus Standard Suction (SS) Strategy for Patients Undergoing Minimally Invasive Lung Resection by VATS or Robotic Approach
Brief Title: A Study to Evaluate Routine Chest Tube Management After Minimally Invasive Lung Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Responsible Party: Principal Investigator, Hiran Fernando, MD, Chief of Thoracic Surgery at Allegheny General Hospital, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-005
Record Dates: First submitted 2021-02-02; First posted 2021-06-04 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either the Low Suction or Standard Suction chest tube management group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Low Suction Strategy of Chest Tube Management (Other)
  Interventions: Other: Low Suction Strategy of Chest Tube Management
- Standard Suction Strategy of Chest Tube Management (Other)
  Interventions: Other: Standard Suction Strategy of Chest Tube Management

INTERVENTIONS:
Other: Low Suction Strategy of Chest Tube Management — A digital chest tube will be set to a low pressure mode (-8mmHg) during recovery after minimally invasive lung resection.
  Arms: Low Suction Strategy of Chest Tube Management
Other: Standard Suction Strategy of Chest Tube Management — A digital chest tube will be to the standard suction mode (-20mmHg) during recovery after minimally invasive lung resection.
  Arms: Standard Suction Strategy of Chest Tube Management

SUMMARY:
Chest tubes are routinely required after surgical procedures for lung cancer. This device is a flexible plastic tube that is inserted through the chest wall to remove air or fluid from around your lungs after surgery for lung cancer. There are two general strategies associated with the clinical management of chest tubes, active and passive suction. If suction is compared to driving a car, active suction is similar to pressing the gas pedal while passive suction is like letting your car move on its own. The suction approach taken by surgeons largely depends on how they were trained and some personal biases and beliefs. However there is no general consensus about which chest tube management strategy is best.

This research aims to compare two settings on a digital drainage system, a low suction (LS) mode - passive suction - and standard suction (ss) mode - active suction. From the data collected, the researchers will analyze whether LS or SS will lead to a better recovery after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are undergoing lobectomy or segmentectomy
2. Patients undergoing wedge resection to diagnose, or as definitive therapy for a lung nodule/cancer.
3. Able to understand and sign consent

Exclusion Criteria:

1. Patients undergoing pneumonectomy or bilobectomy
2. Patients undergoing resection for inflammatory conditions such as aspergillosis
3. Patients undergoing diagnostic wedge resection for interstitial lung disease
4. Patients undergoing redo-VATS or thoracotomy on the same side as current planned resection
5. Patients found to have a "frozen chest" at the time of surgery, requiring extensive adhesiolysis,
6. Patients who are discovered to have metastatic disease during the operation, so that resection is no longer indicated.
7. Patients where a clinical decision to place more than one chest-tube is made

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Duration of air-leak | When the subject arrives to the recovery room directly after surgery, then every 24 hours while admitted to the hospital until air leak resolves (on average, up to 4 days)
  Days

SECONDARY OUTCOMES:
Days from operation to chest tube removal | chest tube placement to chest tube removal on average up to 4 days
  Days
Incidence of prolonged air-leak | Categorial variable: Present or not. Determination of category is measured from onset of air-leak to air-leak resolution or 5 days, whichever comes first.
  Rate of subjects who experience an air-leak which lasts for 5 or more days
Duration of hospital stay | Date of surgery to date of discharge (up to 5 days on average)
  Days/Hours
Impact of suction strategy on patients with high Prolonged Air-Leak Score | duration of study participation which is until chest tube is removed, duration of hospital stay, or 30 days from operation, whichever is longer
  Incidence of PAL based suction strategy
Define cut-off air-leak value where prolonged air-leak is likely to occur, or standard suction strategy is preferable | duration of study participation, which is until the chest-tube is removed, duration of initial hospital stay, or 30 days from operation, whichever is longer
  mL/minute

CONTACTS AND LOCATIONS:
Overall Officials: Hiran Fernando, M.D., Principal Investigator — Allegheny Health Network
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Mayor MA, Khandhar SJ, Chandy J, Fernando HC. Implementing a thoracic enhanced recovery with ambulation after surgery program: key aspects and challenges. J Thorac Dis. 2018 Nov;10(Suppl 32):S3809-S3814. doi: 10.21037/jtd.2018.10.106. PMID 30505568
- [Result] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Result] Cerfolio RJ, Bass C, Katholi CR. Prospective randomized trial compares suction versus water seal for air leaks. Ann Thorac Surg. 2001 May;71(5):1613-7. doi: 10.1016/s0003-4975(01)02474-2. PMID 11383809
- [Result] Marshall MB, Deeb ME, Bleier JI, Kucharczuk JC, Friedberg JS, Kaiser LR, Shrager JB. Suction vs water seal after pulmonary resection: a randomized prospective study. Chest. 2002 Mar;121(3):831-5. doi: 10.1378/chest.121.3.831. PMID 11888968
- [Result] Cerfolio RJ, Bryant AS. The benefits of continuous and digital air leak assessment after elective pulmonary resection: a prospective study. Ann Thorac Surg. 2008 Aug;86(2):396-401. doi: 10.1016/j.athoracsur.2008.04.016. PMID 18640304
- [Result] Pompili C, Detterbeck F, Papagiannopoulos K, Sihoe A, Vachlas K, Maxfield MW, Lim HC, Brunelli A. Multicenter international randomized comparison of objective and subjective outcomes between electronic and traditional chest drainage systems. Ann Thorac Surg. 2014 Aug;98(2):490-6; discussion 496-7. doi: 10.1016/j.athoracsur.2014.03.043. Epub 2014 Jun 4. PMID 24906602
- [Result] Brunelli A, Salati M, Pompili C, Refai M, Sabbatini A. Regulated tailored suction vs regulated seal: a prospective randomized trial on air leak duration. Eur J Cardiothorac Surg. 2013 May;43(5):899-904. doi: 10.1093/ejcts/ezs518. Epub 2012 Sep 28. PMID 23024236
- [Result] Lijkendijk M, Licht PB, Neckelmann K. The Influence of Suction on Chest Drain Duration After Lobectomy Using Electronic Chest Drainage. Ann Thorac Surg. 2019 Jun;107(6):1621-1625. doi: 10.1016/j.athoracsur.2018.12.059. Epub 2019 Feb 8. PMID 30742815
- [Result] Holbek BL, Christensen M, Hansen HJ, Kehlet H, Petersen RH. The effects of low suction on digital drainage devices after lobectomy using video-assisted thoracoscopic surgery: a randomized controlled trialdagger. Eur J Cardiothorac Surg. 2019 Apr 1;55(4):673-681. doi: 10.1093/ejcts/ezy361. PMID 30445572